CLINICAL TRIAL: NCT02007772
Title: Effectiveness of TNI (Nasal High-flow) vs. BiPAP (Biphasic Positive Airway Pressure) in Chronic Global Insufficiency in COPD (Chronic Obstructive Pulmonary Disease) Patients
Brief Title: Effectiveness of TNI vs. BiPAP in Chronic Global Insufficiency in COPD Patients
Acronym: TIBICO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Leipzig (Other)
Collaborators: TNI Medical AG (Industry)
Responsible Party: Principal Investigator, Jens Bräunlich, MD, Dr. Jens Braeunlich, University of Leipzig
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: TIBICO
Record Dates: First submitted 2013-09-16; First posted 2013-12-11 (Estimated); Last update posted 2018-11-15 (Actual); Status verified 2018-11

CONDITIONS: COPD Chronic Obstructive Pulmonary Disease
Keywords: COPD, nHF, BiPAP
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- BiPAP breathing support (Active Comparator): BiPAP is used over a period of 6 weeks (outpatient)
  Interventions: Device: nHF; Device: BiPAP
- nHF / TNI breathing support (Experimental): nasal high-flow is used over a period of 6 weeks (outpatient)
  Interventions: Device: nHF; Device: BiPAP

INTERVENTIONS:
Device: nHF — nasal high-flow is used over a period of 6 weeks (outpatient)
  Other Names: nasal high-flow
Device: BiPAP — BiPAP is used over a period of 6 weeks (outpatient)

SUMMARY:
The purpose of this trial ist to investigate the difference of the efficacy of two systems for breath support in patients with COPD.

DETAILED DESCRIPTION:
The trial consists of 12 weeks of therapy that is divided into two sections. In the first 6-week section patients receive treatment with either TNI or BiPAP and in the second 6-week section treatment is changed. The starting therapy is allocated to the patients via randomisation and should be started directly after the baseline visit.

The treatment and the follow-up period end with the second visit after the second treatment section and the patient decides which device he/she wants to use further.

ELIGIBILITY:
Inclusion Criteria:

* presence of COPD with chronic respiratory global insufficiency
* chronic day-hypercapnia with pCO2 >= 50 mmHg and typical symptoms of ventilatory insufficiency OR patients with exacerbation (after abate of acute symptomatology) with documented hypercapnia >= 50 mmHG on preliminary findings
* age 18 or older
* the patient or caretaker must be able to operate the device after a specific training
* patient must be willing to use the nHF-/BiPAP-device for the whole trial period for at least 5 hours/day
* patient must be able to answer the questionnaires
* written informed consent is obtained

Exclusion Criteria:

* presence of acute respiratory insufficiency
* exacerbation of type I or II in the last 4 weeks
* conservative therapy including long-term oxygen therapy according to GOLD update 2011 is not exhausted
* previous treatment with NIV (non-invasive ventilation) in the last 14 days
* clinical instability or acute illness (e.g. acute myocardial infarction, tachycardial atrial fibrillation)
* signs of cardial decompensation (e.g. edema in the lower limbs, pleural effusion)
* other serious concomitant diseases, the assessment of eligibility is at the discretion of the investigator
* contraindications for NIV
* anamnestic suspicion or proven obstructive sleep apnea (OSA)
* relevant systemic infections, assessment of eligibility is at the discretion of the investigator
* BMI > 30
* other additional pulmonary diseases of other genesis or diseases that affect breathing (e.g. mucoviscidosis, scoliosis, muscular diseases)
* lack of compliance
* participation in other interventional trials at the same time
* pregnant or nursing women
* fertile female patients without effective contraceptive measures during trial participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2011-06; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
difference in capillary CO2 carbon dioxide | Baseline, 6 weeks, 12 weeks
  The primary endpoint is the difference of the capillary pC02 between the treatment with nasal high-flow compared with the baseline value.

SECONDARY OUTCOMES:
difference in absolute change of capillary pCO2 (partial pressure of carbon dioxide ) compared with baseline | Baseline, 6 weeks, 12 weeks
frequency of occurrence of normocapnia after intervention | Baseline, 6 weeks, 12 weeks
  Normocapnia is therefore defined as capillary pCO2 <= 45 mmHg
difference of the relative and absolute change of capillary pCO2 compared with baseline | Baseline, 6 weeks, 12 weeks
difference of the absolute change of SaO2 (arterial oxygen saturation) compared with baseline | Baseline, 6 weeks, 12 weeks
difference of the absolute and relative change of base excess compared with baseline | Baseline, 6 weeks, 12 weeks
difference of the values of base excess after treatment with nHF (nasal high-flow) and of base excess after treatment with BiPAP | baseline, 6 weeks, 12 weeks
difference of the absolute change of HCO3- (hydrogen carbonate / bicarbonate) compared with baseline | baseline, 6 weeks, 12 weeks
difference of HCO3- after treatment with nHF and of HC03- after treatment with BiPAP | baseline, 6 weeks, 12 weeks
difference of P0,1 after treatment with nHF and of P0,1 after treatment with BiPAP | baseline, 6 weeks, 12 weeks
difference of PImax after treatment with nHF and of PImax (maximal inspiratory pressure) after treatment with BiPAP | baseline, 6 weeks, 12 weeks
difference of P0,1/PImax after treatment with nHF and of P0,1/PImax after treatment with BiPAP | baseline, 6 weeks, 12 weeks
difference of the absolute change of the results of the 6-minutes walking test compared with baseline | baseline, 6 weeks, 12 weeks
difference of the absolute change of the disease-specific quality of life compared to baseline | baseline, 6 weeks, 12 weeks
  Quality of life is measured by SGQR (The St George's Respiratory Questionnaire), SRI (Severe Respiratory Insufficiency Questionnaire), a VAS referring to the general health status and the Borg-Scale (CR 10)
frequency of occurrence and type of adverse events under trial therapy (both arms) | baseline, 6 weeks, 12 weeks
difference of the values of user-friendliness of both devices | baseline, 6 weeks, 12 weeks
difference of the time both devices were used | baseline, 6 weeks, 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jens Braeunlich, Dr., Study Chair — Medical Faculty University Leipzig
Locations (14):
- Germany (14):
  - Klinik Donaustauf, Zentrum für Pneumologie, Donaustauf, Bavaria
  - Asklepios Fachkliniken München-Gauting, Klinik für Intensivmedizin und Langzeitbeatmung, Muenchen-Gauting, Bavaria
  - Klinikum Nürnberg Nord, Medizinische Klinik 3, Schwerpunkt Pneumologie, Allergologie, Schlafmedizin, Nuremberg, Bavaria
  - RoMed Klinikum Rosenheim, Medizinische Klinik III, Pneumologie, Rosenheim, Bavaria
  - Marienkrankenhaus Kassel gGmbH, Medizinische Klinik / Pneumologie, Kassel, Hesse
  - Evangelisches Krankenhaus Göttingen-Weende gGmbH, Abteilung für Pneumologie, Bovenden, Lower Saxony
  - Fachkrankenhaus Kloster Grafschaft GmbH, Schlafmedizin & häusliche Beatmung, Schmallenberg, North Rhine-Westphalia
  - Diakonisches Werk Bethanien e.V, Klinik für Pneumologie, Solingen, North Rhine-Westphalia
  - Universitätsklinikum Leipzig, Department für Innere Medizin, Neurologie und Dermatologie, Leipzig, Saxony
  - Zentralklinik Bad Berka GmbH, Klinik für Pneumologie, Bad Berka, Thuringia
  - Evangelisches Krankenhaus Bergisch Gladbach, Pneumologie, Bergisch Gladbach
  - HELIOS Klinikum Emil von Behring, Klinik für Pneumologie, Berlin
  - Asklepios Klinik Harburg, Lungenheilkunde (Pneumologie) im Thoraxzentrum, Sektion Pneumologische Intensiv- u. Beatmungsmedizin, Hamburg
  - Waldburg-Zeil Kliniken, Fachkliniken Wangen, Lungenzentrum Süd-West, Wangen